CLINICAL TRIAL: NCT02941900
Title: PERSONALIZED GENOMIC TESTING FOR MELANOMA: MAXIMIZING COMPREHENSION AND HEALTH OUTCOMES IN SKIN CANCER PATIENTS
Brief Title: Interest and Impact of Skin Cancer Genetic Testing
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1243
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Non-melanoma Skin Cancer (NMSC)
Keywords: Genetic Testing; 16-1243
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva sample

GROUPS / COHORTS (1):
- Non-melanoma skin cancers (NMSCs)
  Interventions: Genetic: MC1R genotyping; Behavioral: MC1R Testing Website; Behavioral: Baseline Survey

INTERVENTIONS:
Genetic: MC1R genotyping
Behavioral: MC1R Testing Website — The website includes three educational modules about genetic testing with corresponding knowledge questions.
Behavioral: Baseline Survey

SUMMARY:
The purpose of this study is to learn whether the patient might be interested in skin cancer genetic testing, and if so, what kinds of thoughts, feelings, and behaviors might result from this testing. Testing for skin cancer risk based on the MC1R gene is not currently used in clinical practice; it will be offered in this study for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English fluent as we do not have the resources to translate all the materials including the website and risk feedback materials into other languages
* Prior history of stage 0, I or II NMSC as per EMR or clinical judgment

Exclusion Criteria:

* Inability to provide meaningful informed consent due to cognitive or psychiatric disability as determined by the judgement of the consenting professional or clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK clinics
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
number of patients interested in MC1R testing | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hay, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT02941900/ICF_000.pdf